CLINICAL TRIAL: NCT06861933
Title: The Effects of Scapulohumeral Rehabilitation on Scapula Kinematics and Upper Extremity Functionality in Individuals With Parkinson's Disease: A Single Blind Randomized Controlled Trial
Brief Title: The Effects of Scapulohumeral Rehabilitation on Scapula Kinematics and Upper Extremity Functionality in Individuals With Parkinson's Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Burdur Mehmet Akif Ersoy University (Other)
Collaborators: Pamukkale University (Other)
Responsible Party: Principal Investigator, Betül Söylemez, Lecturer, PT.MSc., Burdur Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-60116787-020-491421
Record Dates: First submitted 2025-02-26; First posted 2025-03-06 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Parkinson's Disease (PD); Physiotherapy and Rehabilitation
Keywords: Parkinson's Disease; Phsyiotherapy and rehabilitation; upper extremity; neurorehabilitation; scapulahumeral rehabilitation
MeSH Terms: interventions — Physical Therapy Modalities; Rehabilitation; Neurological Rehabilitation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: Scapulohumeral Rehabilitation (Experimental): The scapulohumeral rehabilitation group will receive 20 minutes of scapulohumeral exercises in addition to the 10-minute neurorehabilitation program. Scapulohumeral Exercises: Scapular mobilization, scapular retraction, protraction, elevation in the scapular plane and Proprioceptive Neuromuscular Facilitation (PNF) exercises with the repeated contractions method. The exercises will be applied according to the functional capacities of the individuals in the supine, sitting and standing positions with 10 repetitions at the beginning, without weights, using free weights and resistance bands, and the number of repetitions and sets will be progressed every week. The intervention groups will receive a total of 21 treatment sessions, 3 days a week for 7 weeks.
  Interventions: Other: Physiotherapy and rehabilitation
- Group 2: Upper Extremity Neurorehabilitation (Experimental): In addition to the 10-minute neurorehabilitation program, a 20-minute upper extremity neurorehabilitation exercises and a total of 30 minutes of physiotherapy and rehabilitation program will be applied. Scapular retraction, protraction, elevation movements will be performed in the form of Wand exercises with the help of a stick or cane. Exercises will be progressed by increasing the number of repetitions and sets in supine, sitting and standing positions according to the functional level of the participants. The intervention groups will receive a total of 21 treatment sessions, 3 days a week for 7 weeks.
  Interventions: Other: Physiotherapy and rehabilitation
- Control Group (No Intervention): The control group will consist of healthy volunteers of the same age and gender as individuals diagnosed with Parkinson's disease (PD). The control group will not receive any physiotherapy or rehabilitation program and will only receive relevant assessments to compare with the results of individuals with PD.

INTERVENTIONS:
Other: Physiotherapy and rehabilitation — It is reported in the literature that scapulohumeral rehabilitation applied in primary shoulder pathologies is effective. In neurological diseases, a study was found in which scapulohumeral rehabilitation was applied to individuals diagnosed with stroke and reported that it was effective. However, when the literature was examined, no study was found in which scapulohumeral rehabilitation was applied to individuals diagnosed with PD. Therefore, our aim is to compare the effectiveness of the scapulohumeral rehabilitation program to be applied for shoulder dysfunction, which is thought to be one of the early findings in PD and is reported to be related to other main findings in PD, with the upper extremity neurorehabilitation program.
  Other Names: Physiotherapy; Rehabilitation; neurorehabilitation
  Arms: Group 1: Scapulohumeral Rehabilitation; Group 2: Upper Extremity Neurorehabilitation

SUMMARY:
With this study, individuals diagnosed with PD in Burdur province in Turkey will be provided with a physiotherapy and rehabilitation program for the upper extremity, and it is thought that the treatment received by both groups will have a positive effect on the functionality of the individuals. According to the results of our study, it will be determined whether the scapula kinematics and upper extremity functionality of individuals diagnosed with PD are different from healthy individuals of the same age and gender. After the intervention programs applied to the individuals, it is thought that it will contribute to the physiotherapy and rehabilitation programs of individuals with PD by determining whether the scapulohumeral rehabilitation program is superior to the upper extremity neurorehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* For the intervention group:

  * Having been diagnosed with Parkinson's Disease
  * Being between 1-3 according to the Hoehn & Yahr staging
* For the control group:

  * Being of the same age and gender as the individuals diagnosed with Parkinson's disease included in the study

Exclusion Criteria:

* For the intervention group:

  * Refusing to participate in the study
  * Having a full-thickness rotator cuff muscle rupture
  * Having a history of humerus, clavicle, scapula or shoulder surgery
  * Having a history of humerus, clavicle, scapula or shoulder fracture
  * Having a history of any other disease that may affect the ability to stand independently
* For the control group:

  * Refusing to participate in the study
  * Having a full-thickness rupture of the rotator cuff muscles
  * Having a history of humerus, clavicle, scapula or shoulder surgery
  * Having a history of humerus, clavicle, scapula or shoulder fracture

Study Exclusion Criteria for Volunteers:

* Failure to complete the tests included in the study
* Failure to comply with the study schedule, failure to complete sessions
* Incomplete data
* Failure to attend 3 consecutive sessions
* Voluntary withdrawal

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Scapular Index | From enrollment to the end of treatment at 7 weeks
  It is calculated with the formula (distance between sternal notch - coracoid process / posterolateral angle of acromion - horizontal distance between thoracic spine) x 100.
Pectoralis Minor Index | From enrollment to the end of treatment at 7 weeks
  It is calculated with the formula Pectoralis Minor Index = (Pectoralis Minor Length / Participant's height) x 100.
Lateral Scapular Slide Test | From enrollment to the end of treatment at 7 weeks
  In the Lateral Scapular Slide Test, the distance to the thoracic spinous process corresponding to the inferior angle of the scapula is measured in three different positions: arms relaxed at the sides, hands on the iliac crest, and arm in 90-degree shoulder abduction and full internal rotation. The distances between the two sides are compared. A difference of more than 1.5 cm between the two sides is considered asymmetric.
Box and Block Test | From enrollment to the end of treatment at 7 weeks
  150 small wooden cubes are filled from the box where the patient's hand is to be tested to the box next to it. The patient is asked to throw one cube at a time into the empty box next to it. The number of cubes thrown in 60 seconds is counted. The result gives the score. The test is repeated for both hands.
Upper Extremity Functional Index | From enrollment to the end of treatment at 7 weeks
  It is a scale developed by Stratford et al. in 2001 and consists of twenty activity questions. The person scores between 0-4 according to the difficulty of doing the activity. The lowest score in total is 0, the highest score is 80. Low scores indicate that the person has difficulty doing the activity due to the condition of the upper extremity.
Ultrasound | From enrollment to the end of treatment at 7 weeks
  During the evaluation, the patient will be in a sitting position, with the arm next to the body, the forearm in supination and the elbow in full extension. Supraspinatus muscle thickness measurement will be performed by positioning the probe on the fossa supraspinata of the scapula, perpendicular to the skin, along the muscle fibers. The hyperechogenic bone cortex of the fossa supraspinata will be accepted as the landmark. When the muscle fibers are visualized, the thickness of the supraspinatus muscle will be measured from the level where the muscle is observed to be thickest. For the infraspinatus muscle thickness measurement, the hyperechogenic bone cortex of the fossa infraspinata of the scapula will be accepted as the landmark, and the probe will be placed perpendicular to the skin, along the muscle fibers. After the muscle fibers are visualized, the thickness of the infraspinatus muscle will be measured from the level where the muscle is observed to be thickest.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | From enrollment to the end of treatment at 7 weeks
  VAS is a 10-centimeter (cm) scale where 0 is defined as "no pain" and 10 is defined as "unbearable pain". It is a valid and reliable method for assessing the severity of musculoskeletal pain and is frequently used in clinical studies. In a study conducted on patients with chronic musculoskeletal pain, VAS values less than 3.4 cm were classified as mild pain, VAS values between 3.5 and 7.4 cm were classified as moderate pain, and VAS values greater than 7.5 cm were classified as severe pain. The participants' pain severity will be assessed with VAS for resting and activity conditions.
King's Parkinson's Pain Scale | From enrollment to the end of treatment at 7 weeks
  Consists of 14 items divided into seven different areas. Each item is scored by multiplying the severity (0 [no pain] 3 [very severe pain]) (0 [never] 4 [always]). The areas and score ranges are: musculoskeletal pain (0-12 points); chronic pain (0-24 points); pain associated with fluctuation (0-36 points); night pain (0-24 points); orofacial pain (0-36 points); color change, edema (0-24 points); radicular pain (0-12 points).
Range of Motion | From enrollment to the end of treatment at 7 weeks
  Participants' shoulder flexion, abduction, internal and external rotation movements will be evaluated with a manual goniometer. The angle at which shoulder pain develops in active and passive movements will be recorded.
Scapula Angles | From enrollment to the end of treatment at 7 weeks
  The scapula will be evaluated with the inclinometer in three different positions: at rest, with the shoulder at 45 degrees of flexion and 90 degrees of flexion. The difference between the right and left sides will be compared.
New York Posture Rating Chart | From enrollment to the end of treatment at 7 weeks
  Postural changes in 13 different body segments based on observation are scored as 1 point (marked deviation), 3 points (slight deviation), or 5 points (correct posture). The total score ranges from 13 to 65 points, with higher scores indicating correct/normal postural alignment.
PostureScreen Mobile Smartphone Application | From enrollment to the end of treatment at 7 weeks
  It is an image-based method that takes photographs of individuals in the sagittal and frontal planes. The application calculates postural variables using the individual's anatomical points that are digitally marked depending on the number of variables of interest. This process of digitally marking the points consists of drawing the boundaries of anatomical reference points (pelvic iliac crests, greater trochanter, femoral condyle, and ear lobule) directly on the mobile device screen. Body angles are then calculated. As a result, it provides an output file containing the values of the postural variables and images showing the digitized points and their positions relative to a neutral posture.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Burdur Mehmet Akif Ersoy University, Burdur, Burdur
  - Pamukkale University, Denizli, Denizli

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aktas I, Unlu Ozkan F. Pectoralis minor syndrome. Turk J Phys Med Rehabil. 2022 Nov 22;68(4):447-455. doi: 10.5606/tftrd.2023.12037. eCollection 2022 Dec. PMID 36589355
- [Background] Yu IY, Choo YK, Kim MH, Oh JS. The effects of pressure biofeedback training on infraspinatus muscle activity and muscle thickness. J Electromyogr Kinesiol. 2018 Apr;39:81-88. doi: 10.1016/j.jelekin.2018.01.007. Epub 2018 Jan 31. PMID 29454230
- [Background] Boehm TD, Kirschner S, Mueller T, Sauer U, Gohlke FE. Dynamic ultrasonography of rotator cuff muscles. J Clin Ultrasound. 2005 Jun;33(5):207-13. doi: 10.1002/jcu.20124. PMID 16047388
- [Background] Kretic D, Turk T, Rotim T, Saric G. Reliability of Ultrasound Measurement of Muscle Thickness in Patients with Supraspinatus Tendon Pathology. Acta Clin Croat. 2018 Jun;57(2):335-341. doi: 10.20471/acc.2018.57.02.15. PMID 30431728
- [Background] Moreira R, Teles A, Fialho R et al. Mobile Applications for Assessing Human Posture: A Systematic Literature Review. Electronics. 2020; (8):1196. https://doi.org/10.3390/electronics9081196
- [Background] McRoberts LB, Cloud RM, Black CM. Evaluation of the New York Posture Rating Chart for assessing changes in postural alignment in a garment study. Cloth Text Res J 2013;31:81-96. DOI: 10.1177/0887302X13480558
- [Background] Aytar A, Yuruk ZO, Tuzun EH, Baltaci G, Karatas M, Eker L. The Upper Extremity Functional Index (UEFI): cross-cultural adaptation, reliability, and validity of the Turkish version. J Back Musculoskelet Rehabil. 2015;28(3):489-95. doi: 10.3233/BMR-140545. PMID 25322741
- [Background] Mathiowetz V, Volland G, Kashman N, Weber K. Adult norms for the Box and Block Test of manual dexterity. Am J Occup Ther. 1985 Jun;39(6):386-91. doi: 10.5014/ajot.39.6.386. PMID 3160243
- [Background] Shadmehr A, Azarsa MH, Jalaie S. Inter- and intrarater reliability of modified lateral scapular slide test in healthy athletic men. Biomed Res Int. 2014;2014:384149. doi: 10.1155/2014/384149. Epub 2014 May 13. PMID 24900963
- [Background] Borstad JD, Ludewig PM. The effect of long versus short pectoralis minor resting length on scapular kinematics in healthy individuals. J Orthop Sports Phys Ther. 2005 Apr;35(4):227-38. doi: 10.2519/jospt.2005.35.4.227. PMID 15901124
- [Background] Borstad JD. Resting position variables at the shoulder: evidence to support a posture-impairment association. Phys Ther. 2006 Apr;86(4):549-57. PMID 16579671
- [Background] Chaudhuri KR, Rizos A, Trenkwalder C, Rascol O, Pal S, Martino D, Carroll C, Paviour D, Falup-Pecurariu C, Kessel B, Silverdale M, Todorova A, Sauerbier A, Odin P, Antonini A, Martinez-Martin P; EUROPAR and the IPMDS Non Motor PD Study Group. King's Parkinson's disease pain scale, the first scale for pain in PD: An international validation. Mov Disord. 2015 Oct;30(12):1623-31. doi: 10.1002/mds.26270. Epub 2015 Jun 11. PMID 26096067
- [Background] Boonstra AM, Schiphorst Preuper HR, Balk GA, Stewart RE. Cut-off points for mild, moderate, and severe pain on the visual analogue scale for pain in patients with chronic musculoskeletal pain. Pain. 2014 Dec;155(12):2545-2550. doi: 10.1016/j.pain.2014.09.014. Epub 2014 Sep 17. PMID 25239073
- [Background] Boonstra AM, Schiphorst Preuper HR, Reneman MF, Posthumus JB, Stewart RE. Reliability and validity of the visual analogue scale for disability in patients with chronic musculoskeletal pain. Int J Rehabil Res. 2008 Jun;31(2):165-9. doi: 10.1097/MRR.0b013e3282fc0f93. PMID 18467932